CLINICAL TRIAL: NCT03337477
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate a Potassium Normalization Treatment Regimen Including Sodium Zirconium Cyclosilicate (ENERGIZE)
Brief Title: A Study to Evaluate a Potassium Normalization Treatment Regimen Including Sodium Zirconium Cyclosilicate (ZS) Among Patients With S-K ≥5.8
Acronym: ENERGIZE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D9480C00005; 2017-003955-50 (EudraCT Number)
Record Dates: First submitted 2017-10-23; First posted 2017-11-09 (Actual); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; Insulin; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZS+insulin+glucose (Experimental): ZS will be administered in addition to insulin and glucose. Insulin and glucose is the current standard of care to treat serum potassium ≥5.8mmol/L.
  Interventions: Drug: Sodium Zirconium Cyclosilicate(ZS); Drug: Insulin; Drug: Glucose
- Placebo+insulin+glucose (Placebo Comparator): Placebo will be administered in addition to insulin and glucose. Insulin and glucose is the current standard of care to treat serum potassium ≥5.8mmol/L.
  Interventions: Drug: Placebo; Drug: Insulin; Drug: Glucose

INTERVENTIONS:
Drug: Placebo — Suspension administered orally for a treatment period of 24h. 2 sachets administered up to three times over 10h (at 0, 4 and 10h).
  Arms: Placebo+insulin+glucose
Drug: Sodium Zirconium Cyclosilicate(ZS) — Suspension administered orally for a treatment period of 24h. Single dose contains 2 sachets of ZS 5g. 10g administered up to three times over 10h (at 0, 4 and 10h).
  Other Names: ZS, ZS-9
  Arms: ZS+insulin+glucose
Drug: Insulin — Insulin 0.1 units/kg administered as a bolus or for up to 30 minutes.
  Arms: ZS+insulin+glucose
Drug: Glucose — Glucose 25g administered IV <15 minutes before the insulin.
  Arms: ZS+insulin+glucose
Drug: Insulin — Insulin 0.1 units/kg administered as a bolus or for up to 30 minutes.
  Arms: Placebo+insulin+glucose
Drug: Glucose — Glucose 25g administered IV <15 minutes before the insulin.
  Arms: Placebo+insulin+glucose

SUMMARY:
The study is designed to determine if ZS 10g administered up to three times over 10h added to insulin and glucose in patients presenting with hyperkalemia will prove tolerable and efficacious. Patients will receive ZS or Placebo on top of standard of care treatment with insulin and glucose.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age

Potassium ≥5.8 mmol/L

Exclusion Criteria:

Possible pseudohyperkalaemia

Hyperkalaemia caused by any condition for which a therapy directed against the underlying cause of hyperkalaemia would be a better treatment option than treatment with insulin and glucose.

Dialysis session expected within 4h after randomization

Treated with any therapy intended to lower S-K between arriving at the hospital and randomization during Visit 1.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Peacock, MD, Principal Investigator — Baylor College of Medicine
Locations (21):
- United States (10):
  - Research Site, Montgomery, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Detroit, Michigan
  - Research Site, Royal Oak, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
- Denmark (2):
  - Research Site, Esbjerg
  - Research Site, Herning
- Italy (2):
  - Research Site, Novara
  - Research Site, Piombino
- Russia (7):
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

REFERENCES:
- [Derived] Peacock WF, Rafique Z, Vishnevskiy K, Michelson E, Vishneva E, Zvereva T, Nahra R, Li D, Miller J. Emergency Potassium Normalization Treatment Including Sodium Zirconium Cyclosilicate: A Phase II, Randomized, Double-blind, Placebo-controlled Study (ENERGIZE). Acad Emerg Med. 2020 Jun;27(6):475-486. doi: 10.1111/acem.13954. Epub 2020 Mar 28. PMID 32149451
- See also: CSP_redacted_version — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00005&attachmentIdentifier=9d4cb0ca-d8e0-4b32-a380-d6c3a8ce961e&fileName=D9480C00005_CSP_redacted_version.pdf&versionIdentifier=
- See also: SAP_redacted_version — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00005&attachmentIdentifier=4fc8cb3f-61cc-4138-a7bc-9cffc758a6c2&fileName=D9480C00005_SAP_redacted_version.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in the United States, Russia, Denmark and Italy from 13 February 2018 to 21 December 2018.
Pre-assignment Details: Patients with S-K ≥5.8 mmol/L for whom treatment with insulin and glucose to manage hyperkalaemia has been determined medically appropriate by the Investigator. The study originally recruited patients with S-K ≥6.0 mmol/L; however, this inclusion criterion was updated during CSP Amendment to allow enrolment of patients with S-K ≥5.8 mmol/L.
Groups:
- Sodium Zirconium Cyclosilicate (SZC) 10g: SZC will be administered in addition to insulin and glucose.
- Placebo: Placebo will be administered in addition to insulin and glucose.
Period: Overall Study
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Started (Randomized) | 33 | 37
Completed | 22 | 24
Not Completed | 11 | 13
Not completed — not categorized into the listed ones | 11 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo | Total
Number analyzed (Participants) | 33 | 37 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (12.7) | 56.4 (14.4) | 59.0 (13.8)
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 6 | 11 | 17
  >=50 - <65 years | 11 | 18 | 29
  >=65 years | 16 | 8 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 16
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 22 | 26 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Country
  Participants
    Denmark | 0 | 2 | 2
    Italy | 1 | 1 | 2
    Russia | 13 | 14 | 27
    United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Secondary Outcome: Fraction of Patients Responding to Therapy Defined as: S-K <6.0mmol/L Between 1 and 4h and S-K <5.0mmol/L at 4h; and no Additional Potassium Lowering Therapy From 0 to 4h With Exception of the Initial Insulin Treatment
Description: Additional therapies for hyperkalaemia are 2nd dose of insulin, Beta-agonists, Diuretics, Dialysis, Sodium bicarbonate and Potassium binders when administered with the expressed intent to lower S-K. Patients with any missing potassium value from 1h to 4h inclusive will be treated as non-responders.
Time Frame: Baseline to 4h potassium meansurements.
Population: Full analysis set: all randomized patients. However, patients with no baseline or/and post-baseline data (one patient in each group) were excluded from the analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
Proportion of participants | 0.063 | 0.056

2. Secondary Outcome: The Fraction of Patients Achieving Normokalaemia 1, 2 and 4h After Start of Dosing With SZC/Placebo
Description: Proportion of patients achieving normokalaemia, S-K 3.5-5.0 mmol/L, at 1, 2 and 4h after start of dosing
Time Frame: Baseline to 4h potassium meansurements.
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
Proportion of participants
  1h | 0.156 | 0.139
  2h | 0.125 | 0.056
  4h | 0.063 | 0.056

3. Secondary Outcome: The Fraction of Patients Achieving S-K <5.5mmol/l 1, 2, and 4h After Start of Dosing With SZC/Placebo
Time Frame: Baseline to 4h potassium meansurements.
Population: as for outcome 1
Measure: Number; unit: Proportion of paticipants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
Proportion of paticipants
  1h | 0.313 | 0.306
  2h | 0.375 | 0.167
  4h | 0.156 | 0.139

4. Secondary Outcome: The Fraction of Patients Achieving S-K <6.0mmol/l 1, 2, and 4h After Start of Dosing With SZC/Placebo
Time Frame: Baseline to 4h potassium meansurements.
Population: as for outcome 1
Measure: Number; unit: Proportion of paticipants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
Proportion of paticipants
  1h | 0.656 | 0.611
  2h | 0.625 | 0.472
  4h | 0.469 | 0.361

5. Secondary Outcome: The Fraction of Patients Administered Additional Potassium Lowering Therapy Due to Hyperkalaemia From 0 to 4h.
Description: Additional therapies for hyperkalaemia are 2nd dose of insulin, Beta-agonists, Diuretics, Dialysis, Sodium bicarbonate and Potassium binders when administered with the expressed intent to lower S-K.
Time Frame: Baseline to 4h potassium meansurements.
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
Proportion of participants | 0.156 | 0.306

6. Secondary Outcome: Mean Absolute Change in S-K From Baseline to 1h and 2h After Start of Dosing With SZC/Placebo
Description: The least squares means (LS-means) are derived from a linear regression model of absolute change in S-K at 1h and 2h with the following covariates: treatment group; baseline S-K; time from the start of dosing insulin to the start of dosing SZC/placebo and the dose (units/kg) of the first course of insulin. The 95% CI is associated with LS-Means.
Time Frame: Baseline to 2h potassium measurements.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
mmol/L
  1h | -0.67 [-0.90 to -0.44] | -0.67 [-0.89 to -0.45]
  2h | -0.72 [-0.96 to -0.48] | -0.36 [-0.59 to -0.14]

7. Primary Outcome: Mean Absolute Change in S-K From Baseline Until 4h After Start of Dosing With SZC/Placebo
Description: The least squares means (LS-means) are derived from a linear regression model of absolute change in S-K at 4h with the following covariates: treatment group; baseline S-K; time from the start of dosing insulin to the start of dosing SZC/placebo and the dose (units/kg) of the first course of insulin. The 95% CI is associated with LS-Means.
Time Frame: Baseline to 4h potassium measurements.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g | Placebo
Number analyzed (Participants) | 32 | 36
mmol/L | -0.41 [-0.63 to -0.19] | -0.27 [-0.48 to -0.07]

ADVERSE EVENTS:
Time Frame: AEs, including SAEs, were collected from time of signature of informed consent form throughout the treatment period and including the follow-up period (visit 2 or last contact). AE/SAEs occurring between 0h to 24h and AE/SAEs occurring after 24h (time calculated from the start of the administration of insulin) were analysed separately.
Description: Patients at risk are the ones who got at least one dose, namely 29 in SZC and 33 in placebo.
Groups:
- Sodium Zirconium Cyclosilicate (SZC) 10g (0-24h): SZC will be administered in addition to insulin and glucose. AEs collected between 0-24h.
- Placebo (0-24h): Placebo will be administered in addition to insulin and glucose. AEs collected between 0-24h.
- Sodium Zirconium Cyclosilicate (SZC) 10g (After 24h): SZC will be administered in addition to insulin and glucose. AEs collected after 24h.
- Placebo (After 24 h): Placebo will be administered in addition to insulin and glucose. AEs collected after 24h.
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) 10g (0-24h) | Placebo (0-24h) | Sodium Zirconium Cyclosilicate (SZC) 10g (After 24h) | Placebo (After 24 h)
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/33 | 0/29 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/33 | 2/29 | 3/33
Other Adverse Events (participants affected / at risk) | 4/29 | 5/33 | 3/29 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) 10g (0-24h) (N=29) | Placebo (0-24h) (N=33) | Sodium Zirconium Cyclosilicate (SZC) 10g (After 24h) (N=29) | Placebo (After 24 h) (N=33)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clonic convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Zirconium Cyclosilicate (SZC) 10g (0-24h) (N=29) | Placebo (0-24h) (N=33) | Sodium Zirconium Cyclosilicate (SZC) 10g (After 24h) (N=29) | Placebo (After 24 h) (N=33)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was stopped at 70 patients randomized instead of 132, as initially planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT03337477/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03337477/SAP_001.pdf